CLINICAL TRIAL: NCT03387722
Title: Assessment of Treatment Patterns of Severe Asthmatic Patients Across the Gulf Region - SevEos Study SevEos is a Cross-sectional, Multi-center, Non-interventional Study Aimed to Describe the Treatment Patterns in 250 Severe Asthma Patients Across the Gulf Region.
Brief Title: Assessment of Treatment Patterns of Severe Asthmatic Patients Across the Gulf Region - SevEos Study
Acronym: SevEos
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D2287R00124
Record Dates: First submitted 2017-12-11; First posted 2018-01-02 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Severe Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
SevEos is a cross-sectional, multi-center, non-interventional study aimed to describe the treatment patterns in 250 severe asthma patients across the Gulf region. In addition, the study will determine the current level of asthma control and quality of life in these patients; describe the exacerbation patterns; and determine the current levels of blood eosinophils for the enrolled patients.

DETAILED DESCRIPTION:
The primary objective of this study is to describe the treatments patterns of severe asthmatic patients across four Gulf countries during the past year.

Secondary Objectives

1. To determine the current level of asthma control in these patients. In addition, a comparison of uncontrolled asthma between those with a eosinophilic count ≥ 300 cell/μl and those with an elevated eosinophilic count less than that.
2. To determine the current and past year levels of blood eosinophils, and the percentage of patients with elevated eosinophilic level ≥ 150 cells/μL and ≥ 300 cells/μL
3. To describe the frequency of exacerbations during the past year.
4. To assess the current quality of life (QoL) of these patients.
5. To determine the past year levels of serum IgE.
6. Exploratory objective: To determine the past year levels of other inflammatory biomarkers like periostin and fraction of exhaled nitric oxide (FeNO).

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, patients (both male and female) must fulfill all of the following criteria:

1. Age above 12 years.
2. Body weight of ≥40 kg.
3. Diagnosed by a physician with severe asthma, who requires regular treatment with medium or high dosage Inhaled Corticosteroids (ICS) (patients aged 12-17 years) OR high-dosage ICS ( plus Long-Acting Beta Agonist (LABA) for at least 1 year before enrolment.

[Note that the value of the medium/high dosage is dependent on the type of ICS

Exclusion Criteria:

Patients who meet any of the following criteria are ineligible to participate in the study:

1. Patient refuses to consent.
2. Another clinically important pulmonary disease is considered to be the primary diagnosis, other than severe asthma (i.e.: COPD, major bronchiectasis, active tuberculosis, and other conditions considered by the principal investigator).
3. Mentally disabled patient or inability to understand the study questions.
4. Unable to read/write.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Severe asthma, who requires regular treatment with medium or high dosage Inhaled Corticosteroids (ICS) (patients aged 12-17 years) OR high-dosage ICS ) plus Long-Acting Beta Agonist (LABA) for at least 1 year before enrolment
Sampling Method: Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2017-12-31 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2019-01-03 (Actual)

PRIMARY OUTCOMES:
Asthma treatment and its patterns through generic names. | 1 year
  Changes in Asthma treatment stages during the last year based on the number of prescribed:
  * Short-acting: muscarinic antagonists (SAMA),
  * long-acting muscarinic antagonists (LAMA),
  * Long-acting Beta agonist (LABA),
  * Corticosteroids (Inhaled(ICS), Oral(OCS) & Parental),
  * Theophylline,
  * Biologics.
Asthma treatment and its patterns through dosage | 1 Year
  Changes in Asthma treatment stages during the last year based on the dosage:
  * Short-acting: muscarinic antagonists (SAMA),
  * long-acting muscarinic antagonists (LAMA),
  * Long-acting Beta agonist (LABA),
  * Corticosteroids (Inhaled(ICS), Oral(OCS) & Parental),
  * Theophylline,
  * Biologics.

SECONDARY OUTCOMES:
Asthma Control | 1 year
  Asthma control will be assed using "The Asthma Control Questionnaire". The questionnaire was developed by Elizabeth Juniper( MCSP, MSc Professor, 20 Marcuse Fields) Bosham, West Sussex PO18 8NA, England), to measure both the adequacy of asthma control and change in asthma control, which occurs either spontaneously or as a result of treatment.
  Patients are asked to respond to questions on a 7-point scale (0=no impairment, 6= maximum impairment). The questions are equally weighted and the ACQ score is the mean of the 7 questions and therefore between 0 (totally controlled) and 6 (severely uncontrolled). A change or difference in score of 0.5 is the smallest that can be considered clinically important.
Exacerbations | 1 year
  Collection of exacerbations records based on history of documented Emergency Room(ER),hospital visits and hospitalizations (asthma-related)
quality of life (QoL) | 1 year
  Quality of life will be assed using "Asthma Quality of life Questionnaire with Standardised Activities", a questionnaire developed by Elizabeth Juniper( MCSP, MSc Professor, 20 Marcuse Fields Bosham, West Sussex PO18 8NA, England) to measure the functional problems (physical, emotional, social and occupational) that are most troublesome for patients with asthma. There are 32 questions in the questoinnaire and they are in 4 domains (symptoms, activity limitation, emotional function and environmental stimuli). Patients are asked during the previous two weeks and to respond to 32 questions on a 7-point scale (7 = not impaired at all - 1 = severely impaired). Scores range 1-7, higher scores indicating better quality of life. The better outcome is of higher score value, 0 (totally controlled), 6 (severely uncontrolled).
Eosinophil count | 1 year
  Proportion of severe asthmatics with eosinophil count (threshold ≥150cells/μL and ≥300 cells/μL) based on current/most recent blood eosinophil level during the past year.
level of blood eosinophil. | 1 Year
  Mean or median level of blood eosinophil during the past year.
Total serum IgE | 1 Year
  Mean or median levels of total serum IgE during the past year.
Pre-bronchodilator forced expiratory volume | 1 Year
  Pre-bronchodilator forced expiratory volume in 1 sec
Post-bronchodilator forced expiratory volume | 1 Year
  Post-bronchodilator forced expiratory volume in 1 sec
Pre-bronchodilator expiratory forced vital capacity | 1 Year
  Pre-bronchodilator expiratory forced vital capacity in 1 sec
Post-bronchodilator forced vital capacity | 1 Year
  Post-bronchodilator forced vital capacity in 1 sec

OTHER OUTCOMES:
Periostin level | 1 year
  Mean or median of levels of Last Periostin level during the past year
FeNO level | 1 Year
  Mean or median of levels Last FeNO level during the past year

CONTACTS AND LOCATIONS:
Locations (2):
- Research Site, Muscat, Oman
- Research Site, Dubai, United Arab Emirates

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D2287R00124&attachmentIdentifier=b749bef4-40ff-4a4b-a47f-e7725b7eabfd&fileName=SevEos_D2287R00124_CSR_Final_V1.0_26_March_2020.pdf&versionIdentifier=